CLINICAL TRIAL: NCT04027205
Title: Surgery Versus PhysiothErapist-leD Exercise for Traumatic Tears of the Rotator Cuff: a Multi-site Pilot and Feasibility Randomised Controlled Trial (the SPeEDy Study)
Brief Title: Surgery Versus PhysiothErapist-leD Exercise for Traumatic Tears of the Rotator Cuff
Acronym: SPeEDy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid-19 disruption
Sponsor: Keele University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University Hospitals of Derby and Burton NHS Foundation Trust (Other); University Hospitals, Leicester (Other); Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government); University Hospitals of North Midlands NHS Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Airedale NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG-0292-19-IPCHS
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Rotator Cuff Tear
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist-led exercise (Experimental): Structured and progressive physiotherapist-led exercise programme. Reflective of current guidance for exercise programmes for people with rotator cuff disorders, an individualised programme developed in relation to the participant's specific goals will be prescribed by the physiotherapist and supported over approximately six contact sessions across a 12-week period.
  Interventions: Other: Physiotherapist-led exercise
- Surgical repair (Active Comparator): Surgical repair of the rotator cuff plus usual post-operative rehabilitation.
  Interventions: Procedure: Surgical repair

INTERVENTIONS:
Other: Physiotherapist-led exercise — A programme of physiotherapist-led exercise over approximately 12 weeks.
  Arms: Physiotherapist-led exercise
Procedure: Surgical repair — Surgical repair of the rotator cuff plus usual post-operative rehabilitation
  Arms: Surgical repair

SUMMARY:
The SPeEDy study is a parallel group, pilot and feasibility randomised controlled trial (RCT) with integrated Quintet Recruitment Intervention (QRI) and further qualitative interviews. The study hypothesis is: In adult patients diagnosed with traumatic tears of the rotator cuff, is it feasible to conduct a future, substantive, multi-site RCT to test the hypothesis that physiotherapist-led exercise is not inferior to surgical repair of the rotator cuff in terms of clinical outcomes but is more cost-effective.

DETAILED DESCRIPTION:
Tears of the rotator cuff are a significant cause of shoulder pain. Rates of surgical repair have risen approximately 200% over the last 20 years across Europe and the USA. 9 189 repairs were undertaken in 2015/ 2016 in the NHS. The cost of surgery ranges from £2 897 to £5 593 meaning that direct NHS treatment costs alone are £26.6 to £51.4 million annually.

If a patient is suspected of having a traumatic rotator cuff tear, then guidance from the British Elbow and Shoulder Society and British Orthopaedic Association suggests this is a 'red flag' needing urgent surgical opinion. But, this guidance is open to question. Three randomised controlled trials (RCT) (n = 252) have been synthesised in a systematic review which concluded that surgery is not more effective than conservative care for rotator cuff tears. But, of the 252 patients included, only 40 (16%), were diagnosed with traumatic tears. Hence, there is a dearth of randomised evidence to inform decision-making.

Given uncertainty about the comparative effectiveness of surgery and considering the cost, risk, for example infection, there is an urgent need to carry out high-quality research in this area.

Research Question: In patients diagnosed with traumatic tears of the rotator cuff, is it feasible to conduct a future multicentre RCT to test the hypothesis that physiotherapist-led exercise is not inferior to surgical repair in terms of clinical outcomes but is more cost-effective.

Research Design: Two-arm, parallel group, pilot and feasibility RCT with nested Quintet Recruitment Intervention (QRI) and qualitative interviews.

Setting: Eight NHS hospitals.

Objectives:

1. Determine feasibility of recruiting and retaining patients,
2. Identify barriers and facilitators to recruitment and retention, including patient and clinician equipoise and proportion and reasons for treatment cross-over (reflective of known challenges in surgical RCTs),
3. Estimate the number of potential and willing sites for the future main trial.

Participants: Adults with traumatic tears of the rotator cuff, eligible for surgery.

Intervention/ control: Participants will be allocated on a 1:1 ratio, stratified by tear size to: 1) Structured and progressive physiotherapist-led exercise; 2) Surgical repair and usual post-operative rehabilitation.

Key feasibility outcomes: 1) Numbers of patients screened, eligible, approached, consenting, randomised, and accepting allocation; 2) Rate of retention and follow-up; 3) Feasibility of recruiting participating sites; 4) Participant satisfaction.

Key clinical outcomes: 1) Shoulder pain and function (Oxford Shoulder Score): Quality of life (EQ-5D-5L) at baseline, three, and six months.

Health economic outcomes: Health care resource use and days lost from work over six-months.

Sample size: 76 participants.

Analysis: Analysis will focus on process outcomes (recruitment, retention, and treatment cross-over). Means and confidence intervals of clinical outcomes will be calculated only to inform the sample size calculation for the future main trial.

The QRI will use targeted methods including interviews with clinicians and patients, audio-recording of recruitment appointments and document review to understand and then develop an action plan to optimise recruitment and informed consent. Semi-structured qualitative interviews will explore treatment acceptability and the data will be analysed thematically.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years)
2. Diagnosed with a symptomatic tear of the rotator cuff following a traumatic incident thought to be of sufficient force to induce a tear.
3. Rotator cuff tear confirmed by diagnostic ultrasound or MRI scan undertaken as part of routine diagnostic work-up
4. Eligible for rotator cuff repair surgery or a programme of physiotherapist-led exercise as determined by the attending clinician (surgeon or physiotherapist, where appropriate)
5. Able to return to the participating NHS hospital or associated orthopaedic and physiotherapy services (where physiotherapists have been trained in trial interventions) for post-operative rehabilitation or the programme of physiotherapist-led exercise.
6. Able to understand English.

Exclusion Criteria:

1. Not eligible for rotator cuff repair surgery or a programme of physiotherapist-led exercise as determined by the attending clinician (surgeon or physiotherapist, where appropriate)
2. Patients who are unable to give full informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Numbers of patients screened, number eligible, number approached, number consenting, number randomised, and number accepting allocation | Over recruitment period, 15 months
  Numbers of patients screened, number eligible, number approached, number consenting, number randomised, and number accepting allocation will be recorded descriptively
Numbers of participants continuing in allocated treatment | Six months
  Numbers of participants continuing in allocated treatment will be recorded descriptively
Follow-up response rates to questionnaires (including Oxford Shoulder Score and EQ-5D-5L) | Three months post-randomisation
  Follow-up response rates to questionnaires will be recorded descriptively
Follow-up response rates to questionnaires (including Oxford Shoulder Score and EQ-5D-5L) | Six months post-randomisation
  Follow-up response rates to questionnaires will be recorded descriptively
Determination of zone of clinical equipoise | Over recruitment period, 15 months
  Data from screening logs, including reasons for not approaching potentially eligible patients will be recorded descriptively to inform determination of zone of clinical equipoise
Treatment cross-over | Six months
  Numbers of participants receiving treatment (surgery or PT-led exercise) other than that which was allocated to determine proportion of participants who cross-over will be recorded descriptively
Participant satisfaction with the interventions: five-point ordinal scale | Six months
  Participant satisfaction with the interventions on a five-point ordinal scale; Very Satisfied/Satisfied/Neutral/Dissatisfied/Very Dissatisfied

SECONDARY OUTCOMES:
Pain and disability assessed using the Oxford Shoulder Score (OSS) | Three and six months post-randomisation
  The OSS is a 12-item shoulder-specific self-report measure of shoulder pain and function primarily for the assessment of outcome of shoulder surgery in RCTs. The OSS is reliable, valid, responsive and acceptable to patients. The items refer to the past 4 weeks with five ordinal response options scored from 0 to 4, with 4 representing the best outcome. When the 12 items are summed, this produces an overall score ranging from 0 to 48, with 48 being the best outcome.
Health related quality of life assessed using the EQ-5D-5L | Three and six months post-randomisation
  The EQ-5D-5L is a generic measure of health related quality of life that provides a single index value for health status that can be used for the purpose of clinical and health economic evaluation. The EQ-5D-5L consists of questions relating to five health domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and respondents rate their degree of impairment using five response levels (no problems, slight problems, moderate problems, severe problems and extreme problems). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. A total of 3125 possible health states can be defined in this way which can then be converted in to a single index value between 0 and 1,
Days lost from work due to the shoulder problem | Three and six months post-randomisation
  Days lost from work due to the shoulder problem will be recorded descriptively on a self-report questionnaire
Time taken to return to driving | Three and six months post-randomisation
  Time taken to return to driving will be recorded descriptively on a self-report questionnaire

OTHER OUTCOMES:
Number of recruiting participating sites and numbers of additional sites who are interested in participating in the main trial | Whole study period, 36 months
  Number of recruiting participating sites and numbers of additional sites who are interested in participating in the main trial will be recorded descriptively
Number and type of adverse events | Up to six months post-randomisation
  Number and type of adverse events will be recorded descriptively following patient or clinician report

CONTACTS AND LOCATIONS:
Overall Officials: Chris Littlewood, PhD, Principal Investigator — Manchester Metropolitan University
Locations (1):
- University Hospital of Derby & Burton NHS, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The anonymised datasets generated during and/or analysed during the current study are/will be available upon request from primarycare.datasharing@keele.ac.uk. Core data will be available immediately after publication of the trial results. A data request form is required to be completed and must outline the type of data to be obtained, the reason for obtaining this data (research question / objective), the timing for when the data is required to be available (start date/end date). Checks will be performed by a Data Custodian and Academic Proposals (DCAP) committee at Keele to ensure that the data set requested is appropriately suited to answer the research question/objective and that the request fits with the original ethical approval and participant consent and adheres to funder and legal restrictions. Only de-identified data are available for request in aggregated format or at the level of the individual participant.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Littlewood C, Wade J, Butler-Walley S, Lewis M, Beard D, Rangan A, Bhabra G, Kalogrianitis S, Kelly C, Mehta S, Singh HP, Smith M, Tambe A, Tyler J, Foster NE. Protocol for a multi-site pilot and feasibility randomised controlled trial: Surgery versus PhysiothErapist-leD exercise for traumatic tears of the rotator cuff (the SPeEDy study). Pilot Feasibility Stud. 2021 Jan 7;7(1):17. doi: 10.1186/s40814-020-00714-x. PMID 33413664
- [Derived] Littlewood C, Astbury C, Bush H, Gibson J, Lalande S, Miller C, Pitt L, Tunnicliffe H, Winstanley R. Development of a physiotherapist-led exercise programme for traumatic tears of the rotator cuff for the SPeEDy study. Physiotherapy. 2021 Jun;111:66-73. doi: 10.1016/j.physio.2020.07.008. Epub 2020 Aug 3. PMID 33316867

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT04027205/Prot_SAP_000.pdf